CLINICAL TRIAL: NCT02253615
Title: Effects of 16 Weeks of Resistance Training Using Elastic Resistance or Machines on Muscle Mass, Strength and Postural Control in Untrained Older Adults.
Brief Title: Effects of Resistance Training in Untrained Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Wagner Rodrigues Martins, PhD, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERT-2014
Record Dates: First submitted 2014-09-25; First posted 2014-10-01 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Aging; Older Adults
Keywords: Aging; Resistance training; Muscle strength; Functional performance; Postural balance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Machine resistance training (MRT) (Active Comparator): The machine resistance training will consist of four exercises for lower limbs and four exercises for upper limbs which will be alternately performed with a one-minute interval between them during familiarization and training periods. Lower limb exercises will consist of: hip extension and abduction, and knee flexion and extension. Upper limb exercises will consist of: bench press, rowing, triceps and high pulley exercise.
  Interventions: Other: Machines exercises
- Elastic resistance training (ERT) (Experimental): The elastic resistance training will consist of four exercises for lower limbs and four exercises for upper limbs which will be alternately performed with a one-minute interval between them during familiarization and training periods. Lower limb exercises will consist of: hip extension and abduction, and knee flexion and extension. Upper limb exercises will consist of: bench press, rowing, triceps and high pulley exercise.
  Interventions: Other: Elastic exercises

INTERVENTIONS:
Other: Machines exercises — Resistance training in pneumatic machines.
  Arms: Machine resistance training (MRT)
Other: Elastic exercises — Resistance training with elastic tubes.
  Arms: Elastic resistance training (ERT)

SUMMARY:
The latest randomized controlled trials and systematic reviews of resistance training performed by older adults reported that the systematic use of exercise in machines improves muscle strength and power, functional abilities, body mass and body balance. However, the effect of resistance training with elastic tubes exercises have not been studied in all the variables described above. The objective of this study is to analyze the effects of elastic tubes exercises on muscle mass, muscle strength, functional performance and postural control in elderly untrained.

DETAILED DESCRIPTION:
This is a randomized clinical trial study (RCT) with 2 parallel arms. The subjects will be divided in 2 groups with a randomized block technique: Elastic Training Group (ETG) and Machine Training Group (MTG). The subjects will be submitted to a two-week familiarization period and then a sixteen-week of strength training program will be performed twice a week.

This regimen of resistance training in both groups will consist of four exercises for lower limbs and four exercises for upper limbs which will be alternately performed with a one-minute interval between them during familiarization and training periods. Lower limb exercises will consist of: hip extension and abduction, and knee flexion and extension. Upper limb exercises will consist of: bench press, rowing, triceps and high pulley exercise.

ELIGIBILITY:
Inclusion Criteria:

* Convenience sample of forty healthy older adults with a minimum of 55 years of age.

Exclusion Criteria:

* subjects suffering from orthopedic, neurologic, rheumatologic, metabolic or heart conditions, and uncontrolled arterial hypertension. Additional exclusion criteria included undergoing estrogen therapy, use of cardiac pacemaker, knee or hip arthroplasty, the presence of fragments from previous osteosynthesis; orthopedic surgery, fractures, muscle injury or the practice of resistance training within the last 6 months

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass | Change from baseline in body mass at 16 weeks.
  To assess muscle mass, a Dual-energy X-ray Absortiometry (DXA) (GE Electric Company®, Lunar Prodigy) will be used.
Change in Muscle Strength | Change from baseline in muscle strength at 16 weeks.
  Lower limb muscle strength will be assessed with an isokinetic dynamometer (Biodex System®, model III) and upper limb muscle strength with an isometric dynamometer (Jamar®, Hand Dynamometer).
Change in Postural Balance | Change from baseline in postural balance at 16 weeks.
  The postural balance will be assessed with a three-dimensional (3D) motion analysis system and force plates.

SECONDARY OUTCOMES:
Change in Functional performance | Before and after 16 weeks of resistance training
  The functional performance will be assessed with Ten Meters Walk Test (TMW), Timed Up&Go Test (TUG) and 30 Second Chair Stand Test (T30).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Brasilia, Brasília, Federal District, Brazil

REFERENCES:
- [Background] Lorenz DS. Variable resistance training using elastic bands to enhance lower extremity strengthening. Int J Sports Phys Ther. 2014 May;9(3):410-4. PMID 24944861
- [Background] Joy JM, Lowery RP, Oliveira de Souza E, Wilson JM. Elastic Bands as a Component of Periodized Resistance Training. J Strength Cond Res. 2016 Aug;30(8):2100-6. doi: 10.1519/JSC.0b013e3182986bef. PMID 23669815
- [Background] Martins WR, de Oliveira RJ, Carvalho RS, de Oliveira Damasceno V, da Silva VZ, Silva MS. Elastic resistance training to increase muscle strength in elderly: a systematic review with meta-analysis. Arch Gerontol Geriatr. 2013 Jul-Aug;57(1):8-15. doi: 10.1016/j.archger.2013.03.002. Epub 2013 Apr 4. PMID 23562413
- [Result] American College of Sports Medicine; Chodzko-Zajko WJ, Proctor DN, Fiatarone Singh MA, Minson CT, Nigg CR, Salem GJ, Skinner JS. American College of Sports Medicine position stand. Exercise and physical activity for older adults. Med Sci Sports Exerc. 2009 Jul;41(7):1510-30. doi: 10.1249/MSS.0b013e3181a0c95c. PMID 19516148
- [Result] Colado JC, Garcia-Masso X, Pellicer M, Alakhdar Y, Benavent J, Cabeza-Ruiz R. A comparison of elastic tubing and isotonic resistance exercises. Int J Sports Med. 2010 Nov;31(11):810-7. doi: 10.1055/s-0030-1262808. Epub 2010 Aug 11. PMID 20703977
- [Derived] Martins WR, Safons MP, Bottaro M, Blasczyk JC, Diniz LR, Fonseca RM, Bonini-Rocha AC, de Oliveira RJ. Effects of short term elastic resistance training on muscle mass and strength in untrained older adults: a randomized clinical trial. BMC Geriatr. 2015 Aug 12;15:99. doi: 10.1186/s12877-015-0101-5. PMID 26265075